CLINICAL TRIAL: NCT03837665
Title: Efficacy of Platelet Enriched Plasma in Preventing Surgery for Patients With Chronic Tympanic Membrane Perforation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment barriers
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Hinrich Staecker, MD, PhD, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00140843
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Tympanic Membrane Perforation
Keywords: Platelet Rich Plasma; TM perforations; Hearing loss; Hole in the eardrum
MeSH Terms: conditions — Tympanic Membrane Perforation; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP Treatment (Experimental): Participants receive platelet rich plasma treatment. Participants will be asked to make up to 5 trips to the clinic (one for eligibility, one for the PRP, three follow-up visits). Participation is expected to last up to about 6 weeks. After the second visit and application of PRP, patients will be monitored closely for any complications or concerns. This will include a follow up phone call 3-5 days after the initial application of PRP. Patients will also be followed closely in 2 week intervals or sooner should any problems or concerns arise.
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Platelet Rich Plasma (PRP) is blood plasma that has been enriched with platelets.
  Other Names: PRP

SUMMARY:
By doing this study, researchers hope to find out if platelet rich plasma (PRP) can heal holes in the eardrum as an alternative to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet criteria for tympanoplasty procedure
* Willing to comply with the protocol and attend all study visits
* Able to provide written informed consent

Exclusion Criteria:

* Patients who have previously undergone middle ear or lateral skull base surgery
* Patients who would not qualify for a tympanoplasty
* Any type of platelet disorder, cancer, or ongoing systemic infection
* Any type of hemodynamic instability, septicemia, infection, tobacco use, any use of steroids to the ear drums
* Type I diabetes or other autoimmune pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hinrich Staecker, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRP Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 0 participants reported because only 1 participant was enrolled and therefore confidentiality is an issue.
Arm/Group | PRP Treatment
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Patients Requiring Surgery
Description: Number of participants that are able to avoid surgery for their perforation.
Time Frame: 6 Weeks
Population: 0 participants reported because only 1 participant was enrolled and therefore confidentiality is an issue.
Arm/Group | PRP Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Healing
Description: Size of perforation
Time Frame: 6 Weeks
Population: 0 participants reported because only 1 participant was enrolled and therefore confidentiality is an issue.
Arm/Group | PRP Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | PRP Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT03837665/Prot_SAP_000.pdf